CLINICAL TRIAL: NCT05806801
Title: Metabolic Adaptations to Weight Loss With and Without Exercise
Acronym: WAX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Professor of Movement Science and Director of the Substrate Metabolism Laboratory (SML) at the University of Michigan School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00220220
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Metabolic Disease; Metabolic Syndrome; Insulin Sensitivity; Insulin Resistance; Weight Loss
MeSH Terms: conditions — Obesity; Metabolic Diseases; Metabolic Syndrome; Insulin Resistance; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate Intensity Continuous Training (MICT) exercise group (Experimental): 45 minutes of continuous steady-state exercise at 70% maximal heart rate throughout the 10% weight loss phase of the study
  Interventions: Behavioral: MICT Exercise
- No exercise (Control) (Experimental): to remain sedentary (no planned physical exercise) throughout the duration of the 10% weight loss phase of the study
  Interventions: Behavioral: No Exercise (Control)

INTERVENTIONS:
Behavioral: MICT Exercise — Subjects randomized into this group will complete a moderate intensity continuous exercise 4 days/week.
  Arms: Moderate Intensity Continuous Training (MICT) exercise group
Behavioral: No Exercise (Control) — Subjects randomized into this group will remain sedentary throughout the duration of the study.
  Arms: No exercise (Control)

SUMMARY:
Study Purpose:

The combination of caloric restriction and exercise is the most common first-line treatment for obesity-related disorders, yet we know very little about how these two very different treatments work together. A deeper understanding about mechanisms underlying the health benefits of adding exercise to a weight loss program will not only aid efforts to optimize more effective lifestyle interventions, but it can also uncover novel targets for the treatment/prevention of obesity-related diseases.

Although a reduction in body fat is the fundamental adaptation to weight loss, we know almost nothing about the effects that adding exercise has on structural and functional changes within fat tissue that may further enhance metabolic health. This is very important because many obesity-related metabolic health complications are tightly linked with abnormalities in abdominal fat tissue. We argue exercise-induced modifications in abdominal fat tissue will reveal persistent health benefits even if some weight is regained

Study Summary:

10% Weight Loss Phase - Subject participation in the study will involve a series of metabolic tests before, at midpoint, and after undergoing a 10% weight loss program (with or without exercise training depending on group randomization). During this, subjects will be randomized into one of two different experimental groups:

1. Moderate Intensity Continuous Training (MICT) exercise group
2. No exercise (control) group

Follow-up Phase: After completing the metabolic testing post-weight loss, all study-related diet and exercise supervision will end and subjects will be free to make their own choices regarding diet and exercise/physical activity behavior. Subjects will then be asked to complete follow-up testing at 2-, 4- and 6- months post-weight loss.

Total involvement in the study for each subject will likely be about 10-13 months (4-7 months during weight loss phase, 6 months during follow-up phase).

ELIGIBILITY:
Inclusion criteria

* Age: 18-40
* Body Mass Index: 30-40 kg/m2
* Weight stable (±3kg for greater than or equal to about 2 months)
* No regularly planned exercise/physical activity
* Women must have regularly occurring menses and must be premenopausal

Exclusion criteria

* EKG abnormalities
* Evidence/history of cardiovascular disease, diabetes or other metabolic disease
* Medications known to affect lipid or glucose metabolism
* Pregnant or lactating
* Tobacco or e-cigarette use
* Prior experience of hypersensitivity to insulin, human albumin, and potassium chloride injection.
* Allergies/hypersensitivity to local anesthetics of the amide type (e.g., lidocaine)
* History of hyperkalemia or potential for developing hyperkalemia (including but not limited to taking drugs that may induce hyperkalemia such as cardiac glycosides or potassium sparing diuretics)
* Anti-coagulant medication (e.g., Coumadin, Rivaroxaban) and Lidocaine allergy/sensitivity are exclusion criteria for the biopsy procedure.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 2 hours
  a hyperinsulinemic-euglycemic clamp will be used to quantify peripheral insulin sensitivity
Fatty acid turnover | 2 hours
  stable isotope tracer infusion methods will be used to assess fatty acid turnover
Adipose tissue capillarization | 30 minutes
  measured immunohistochemically using an antibody for CD31, quantified using ImageJ software
Adipose tissue fibrosis | 30 minutes
  measured histologically using Sirus Red Staining, quantified using ImageJ software

SECONDARY OUTCOMES:
Body weight change | 6 months
  Change in body weight will be assessed 6 months after completing the 10% weight loss intervention
Body fat mass | 30 minutes
  Body fat mass will be measured by Dual Energy X-ray Absorptiometry (DEXA)
Oral Glucose Tolerance Test (OGTT) | 2 hours
  A test in which glucose is given and blood samples taken afterward to determine how quickly it is cleared from the blood will be completed at each clinical visit appointment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Horowitz, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No